CLINICAL TRIAL: NCT05898347
Title: Nevoid Basal Cell Carcinomas in Young People With Gorlin Syndrome
Brief Title: Nevoid Basal Cell Carcinomas in Gorlin Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kristin Halvorsen Hortemo, Associate Professor, Medical Doctor, Oslo University Hospital
Other Study IDs: 487620
Record Dates: First submitted 2023-05-29; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Basal Cell Carcinoma; Gorlin Syndrome
Keywords: Dermatoscopy
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gorlin syndrome: Children aged six to seventeen years old with Gorlin syndrome and nevoid basal cell carcinomas.
  Interventions: Other: Active surveillance

INTERVENTIONS:
Other: Active surveillance — Skin lesions clinically compatible with nevoid basal cell carcinomas are documented with measurements, clinical description, clinical photos and dermatoscopy photos every eight months for two years. Three representative skin lesions are selected at the first visit to be removed by skin biopsy at the end of the observation period (two years) for histopathological analyses.
  If a nevoid basal cell carcinoma shows a certain increases in size (according to pre-specified criteria of the study protocol), ulcerates, gets unevenly demarcated or give functional complaints during the observation period, the skin lesion will be excised.

SUMMARY:
The overall aim of the project is to gain knowledge about the expected course of nevoid basal cell carcinomas and the usefulness of dermatoscopy in young individuals with Gorlin syndrome.

Clinical experience and some case-reports suggest that nevoid basal cell carcinomas have an indolent course with slow growth and that they can sometimes regress. However, no systematic research has previously been performed.

Increased knowledge about nevoid basal cell carcinomas and the use of dermatoscopy could be of great clinical value in the follow-up and treatment of individuals with nevoid basal cell carcinoma syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The individual has Gorlin syndrome (clinically and/or genetically diagnosed)
* The individual is minimum 6 years and maximum 17 years
* The individual has at least three skin lesions clinically compatible with nevoid basal cell carcinomas

Exclusion Criteria:

* The patient has a psychiatric disorder not compatible with completion of the study examinations
* The patient has received topical treatment (imiquimod, 5-fluorouracil, photodynamic therapy and/or cryotherapy) of nevoid basal cell carcinomas during the last three months

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged six to seventeen years with Gorlin syndrome and nevoid basal cell carcinomas living in Norway.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nevoid basal cell carcinoma size increase | Two years
  Largest diameter (measured in millimeter) of nevoid basal cell carcinomas after two years surveillance compared to at baseline.
Dermatoscopy findings | Two years
  Dermatoscopy findings of nevoid basal cell carcinomas compared to nevoid basal cell carcinoma size increase.

SECONDARY OUTCOMES:
Nevoid basal cell carcinoma histology | Two years
  Histological analysis, including immune histochemistry, of skin biopsies obtained from representative nevoid basal cell carcinomas.

OTHER OUTCOMES:
Clinical manifestations associated with nevoid basal cell carcinomas | Two years
  Presence of congenital anomalities and benign neoplasias (odontogenic keratocysts, other cysts, fibromas) in patients with nevoid basal cell carcinomas.
Mutation burden in nevoid basal cell carcinomas analyzed by next-generation sequencing | Two years
  Next-generation sequencing of DNA extracted from skin biopsies obtained from representative nevoid basal cell carcinomas, including genes described in skin carcinomas.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Hortemo, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway